CLINICAL TRIAL: NCT03667261
Title: Alveolar and Soft Tissue Changes Surrounding Immediate Implant in the Mandibular Molars With and Without Using Sealing Socket Abutment Technique (Randomized Clinical Trial)
Brief Title: Using Sealing Socket Abutment Technique With Immediate Implant in the Mandibular Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Amen Zahran, clinical research, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01118111027
Record Dates: First submitted 2018-07-18; First posted 2018-09-12 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Soft Tissue Mass

STUDY DESIGN:
Intervention Model Description: cases with with hopeless mandibular molars followed by immediate implant placement
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blinded as well as the data analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cover screw (Active Comparator): extraction of hopeless mandibular molars followed by immediate implants that will be covered using cover screw
  Interventions: Device: cover screw
- sealing socket abutment (Experimental): extraction of hopeless mandibular molars followed by immediate implants that will be covered using sealing socket abutment
  Interventions: Device: Sealing Socket Abutment

INTERVENTIONS:
Device: Sealing Socket Abutment — Sealing Socket Abutment (SSA) serves as a mechanical barrier to isolate the grafted area, stabilize the clot and contain the graft material, and seal the socket from foreign contaminants and also minimizing the risk of premature loading of the implant during healing. By preparing an SSA fabricated to follow the transmucosal contours of the natural tooth, the grafted area can be sealed and separated from the growth of soft tissue without the use of a membrane or releasing incisions
  Other Names: Anatomic Harmony Abutment
  Arms: sealing socket abutment
Device: cover screw — immediate implant placement in mandibular molar area will be covered with conventional cover screw
  Arms: cover screw

SUMMARY:
First and second molar locations present major challenges when immediate implant placement is planned due to large extraction sockets that are difficult to seal without mucoperiosteal flap reflection which is less comfortable to patient and also crestal socket morphology not amenable to standard healing abutment which have circular shape and the possibility of high occlusal forces during function with complete provisional crown.Immediate implant placement without sealing socket abutment has several drawbacks, such as collapse of existing soft tissue and also it needs second stage surgery which is less comfortable to patient and chair time consuming for the operator.

DETAILED DESCRIPTION:
The anatomical changes that occur with the alveolar ridge after the loss of tooth can be a challenge to redevelop during the restorative process. The preservation of the soft tissue level from the time of extraction may optimize the final prosthetic outcome. One technique that can be used to achieve ideal tissue form is immediate dental implant placement with a custom-healing abutment.

Immediate implant placement followed by immediate provisional restoration of single sites is a protocol used to replace a failing tooth. This technique may benefit patients with a thin periodontal biotype. Another benefit is the simplification of the final restorative procedure. Pre-fabricated healing abutments are circular in shape. Attempts at molding the tissue from a small opening above the implant to a contour similar to the missing tooth can take time. The preserved tissue profile can be easily duplicated in the impression process and allow for an accurate fabrication of a restoration in harmony with ideal tissue architecture at the day of insertion.

This form of maintenance of the supporting gingival tissue has been demonstrated to be beneficial using immediate pontics for tooth replacement. Preservation of form, rather than re-creation, is achieved with the extension of the pontic into the subgingival zone with a contour replicating that of the extracted tooth. Concepts from immediate pontics have been applied to immediate dental implants with a similar goal. This is achieved with either a custom healing abutment or a complete provisional crown. The use of a custom-healing abutment is recommended in patients who have a deep anterior bite, who present with signs of bruxism, or who have a malocclusion that is not conducive to the protection of an immediate restoration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hopeless molars in the posterior area of the mandible.
* Both sexes.
* No intraoral soft and hard tissue pathology
* No systemic condition that contraindicate implant placement

Exclusion Criteria:

* Very thin less than 0.5 mm or absent buccal plate.
* Heavy smokers more than 10 cigarettes per day.
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems
* Disorders to implant are related to history of radiation therapy to the head and neck neoplasia, or bone augmentation to implant site
* Immunodeficiency pathology, bruxism, stress situation (socially or professionally), emotional instability, and unrealistic aesthetic demands.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Soft tissue changes around implant | 18 months
  The PES comprises the following five variables: mesial papilla, distal papilla, curvature of the facial mucosa, level of the facial mucosa, and root convexity/soft tissue, color and texture at the facial aspect of the site. Using a 0-1-2 scoring system, 0 being the lowest, 2 being the highest value, the maximum achievable PES is 14 at time of surgery and at the time of final prothesis.
  All ten parameters are assessed by direct comparison with the contralateral tooth and a score of 2, 1, or 0 is assigned to all ten parameters. Thus, a maximum total PES of 10 can be reached which represents the optimum condition of the soft tissues of the rehabilitated site compared to the characteristics of the contralateral natural tooth.

SECONDARY OUTCOMES:
marginal bone loss | 18 months
  The marginal bone on the buccal and lingual surface of the dental implant cannot be assessed with periapical views in millimeters from fixed point .
  Using the same exposure parameter settings selected after a pilot test and images reconstructed with the same slice thickness and a cutting direction for histological matching to compare preoperative and postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: mohamed atef, Principal Investigator — Cairo University
Locations (1):
- Cairo Universty, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided